CLINICAL TRIAL: NCT03099395
Title: Pattern of Repeat Cardiovascular Events During Follow-up After First Diagnosed Event-MI - PRECLUDE-MI - A Retrospective Cohort Study
Brief Title: Pattern of Repeat Cardiovascular Events During Follow-up After First Diagnosed Event-MI
Acronym: PRECLUDE-MI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Uppsala University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: PRECLUDE-MI
Record Dates: First submitted 2017-03-28; First posted 2017-04-04 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Myocardial Infarction
Keywords: myocardial infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No re-MI, one re-MI, > one re-MI: From a population with MI surviving one year (78 468 pts) the number of pts with no re-MI, one re-MI or > re-MI will be described.

SUMMARY:
Recurrent myocardial infarctions (reinfarctions) can be due to recurrence at the original treatment site, the presence of untreated lesions elsewhere, or in progressive lesions. There are scarce published data describing the localization (affected vessel/s) and severity (NSTE-ACS/STE-ACS) of reinfarction(s) compared to the index MI (e.g proportion of recurrent infarctions in the previously diseased vessel) in large unselected patient populations. If reinfarctions are generally more severe than index MI/recurrent MI(s), this might have implications for choice of treatment and treatment length.

Moreover, data from unselected patient populations on the overall incidence pattern/rate of patients experiencing multiple reinfarctions is sparse. Patients who experience multiple ischemic events may be a subset of patients who are poor responders to therapy. There is also a possibility that patients with multiple events are less likely to have received evidence-based therapy such as coronary stenting, novel and more effective antithrombotics and modern lipid lowering treatment for the initial event. Poor adherence to secondary prevention measures (e.g. low compliance to medication and adherence to cardiac rehabilitation programs) may also increase the risk of recurrent events.

Therefore identification of the baseline characteristics, including treatment decision strategies in the setting of a myocardial infarction, among such subjects may allow modifications of the clinical management strategy prior to the occurrence of subsequent ischemic events. Such modifications could include providing a more intensive or additional therapy in certain patient groups or find strategies to improve patient adherence and drug compliance.

A patient with reinfarctions requires more hospitalizations, treatments, laboratory tests, and out-patient visits, resulting in overall increased costs. From the patient perspective, recurrent events result in higher mortality and worsened quality of life.

DETAILED DESCRIPTION:
This study will combine the SWEDEHEART registries RIKS-HIA (Registry of Information and Knowledge about Swedish Heart Intensive care Admissions), SCAAR (Swedish Coronary Angiography and Angioplasty Registry) and SEPHIA (the registry for secondary prevention following coronary intensive care); and the Swedish National Population Registry (to obtain data regarding vital status and date of death), Swedish Cause of Death Register (to separate fatal from non-fatal MI), the Swedish Patient Registry (to obtain data on prior medical history) and the Swedish Drug Registry (to obtain prescribed medical treatment and filled prescriptions).

The RIKS-HIA database covers all acute coronary syndrome (ACS) patients treated at heart intensive care units in Sweden and SCAAR entails all PCI procedures performed across all centers in Sweden.

In this study the investigators will include patients with first time ever of NSTE-ACS and STE-ACS and receiving care at cardiac intensive care units and entered in the SWEDEHEART registry between 1 July 2006 and 31 December 2014. Baseline and in-hospital characteristics will be obtained, including peri-procedural anti-thrombotic treatments.

To assess the incidence rate and fatality of reinfarctions in a contemporary unselected MI cohort

To characterize patients with one and multiple reinfarctions during the observation period vs. those without.

To characterize patients with one and multiple reinfarction during the observational period vs. those without.

ELIGIBILITY:
Inclusion Criteria:

* Patients registered in SWEDHEART with an index-MI within the observation period

Exclusion Criteria:

* Less than one year follow-up data
* Previous MI

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients registered in SWEDHEART with an index-MI within the observation period.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2017-10-01 (Estimated); Study Completion 2017-10-01 (Estimated)

PRIMARY OUTCOMES:
Pattern of repeat cardiovascular events during follow-up after first diagnosed event-MI. | max 8 years follow-up

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Varenhorst C, Hasvold P, Johansson S, Janzon M, Albertsson P, Leosdottir M, Hambraeus K, James S, Jernberg T, Svennblad B, Lagerqvist B. Culprit and Nonculprit Recurrent Ischemic Events in Patients With Myocardial Infarction: Data From SWEDEHEART (Swedish Web System for Enhancement and Development of Evidence-Based Care in Heart Disease Evaluated According to Recommended Therapies). J Am Heart Assoc. 2018 Jan 9;7(1):e007174. doi: 10.1161/JAHA.117.007174. Epub 2018 Jan 4. PMID 31913732